CLINICAL TRIAL: NCT01193517
Title: Phase I/II Study of Azacitidine and CAPOX (Capecitabine + Oxaliplatin) in Metastatic Colorectal Cancer Patients Enriched for Hypermethylation of CpG Promoter Islands
Brief Title: Azacitidine and CAPOX in Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0625; NCI-2010-01973 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-08-31; First posted 2010-09-02 (Estimated); Results first posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Colorectal Cancer
Keywords: Refractory metastatic colorectal cancer; CRC; colorectal adenocarcinoma with metastatic disease; Azacitidine; 5-Azacytidine; 5-aza; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816; Capecitabine; Oxaliplatin; CAPOX; Xeloda; Eloxatin; Hypermethylation; CpG island methylator phenotype
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Azacitidine; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase I (Experimental): Dose Escalation of Azacitidine + CAPOX (Capecitabine, Oxaliplatin)
  Interventions: Drug: Azacitidine; Drug: Capecitabine; Drug: Oxaliplatin
- Phase II (Experimental): MTD of Azacitidine + CAPOX
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Drug: Azacitidine MTD

INTERVENTIONS:
Drug: Azacitidine — Starting dose level 75 mg/m2/day subcutaneously on Days 1-5 of a 21 day cycle.
  Other Names: 5-Azacytidine; 5-aza; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816
  Arms: Phase I
Drug: Capecitabine — 1500 mg/m2/day by mouth twice daily in divided doses on Days 1-14 of a 21 day cycle.
  Other Names: Xeloda
Drug: Oxaliplatin — Starting dose level 90 mg/m2 by vein on Day 2 of a 21 day cycle.
  Other Names: Eloxatin
Drug: Azacitidine MTD — Highest tolerable dose of combination azacitidine with CAPOX found in Phase I.
  Other Names: 5-Azacytidine; 5-aza; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816
  Arms: Phase II

SUMMARY:
The goal of the Phase I portion of this study is to find the highest tolerable dose of azacitidine combined with capecitabine and oxaliplatin (CAPOX) that can be given to patients with metastatic colorectal cancer.

The goal of the Phase II portion of this study is to learn if azacitidine, given in combination with CAPOX, can help to control metastatic colorectal cancer. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Azacitidine is designed to block certain proteins in cancer cells whose job is to stop the function of the tumor-fighting proteins. By blocking the "bad" proteins, the tumor-fighting genes may be able to work better.

Capecitabine is designed to interfere with the growth of cancer cells.

Oxaliplatin is designed to keep new cancer cells from growing.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you joined this study. Up to 4 groups of up to 3-6 participants will be enrolled in the Phase I portion of the study, and up to 30 participants will be enrolled in Phase II.

If you are enrolled in the Phase I portion, the dose of azacitidine and oxaliplatin you receive will depend on when you joined this study. All participants will receive the same dose of capecitabine. The first group of participants will receive a low dose level of the combination. Each new group will receive a higher dose of the combination than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of the combination of azacitidine, oxaliplatin, and capecitabine is found.

If you are enrolled in the Phase II portion, you will receive the combination of azacitidine, oxaliplatin, and capecitabine at the highest dose that was tolerated in the Phase I portion.

Central Venous Catheter (CVC):

Before you can begin to receive oxaliplatin on this study, you will have a CVC placed if you do not have one already. A CVC is a sterile, flexible tube that will be placed into a large vein while you are under local anesthesia. Your doctor will explain this procedure to you in more detail, and you will be required to sign a separate consent form for this procedure.

Study Drug Administration:

A cycle of treatment is defined as 21 days.

Azacitidine will be injected under your skin on Days 1-5 of each cycle.

You will receive oxaliplatin by vein over 2 hours on Day 2 of each cycle.

You will take capecitabine by mouth 2 times each day on Days 1-14 of each cycle. Capecitabine tablets should be taken 12 hours apart, within 30 minutes after eating a meal.

Study Visits:

Up to 3 days before or on Day 1 of each cycle, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight and vital signs.
* You will have a neurosensory assessment.
* Your performance status will be recorded.
* You will be asked about any symptoms and/or side effects you may be experiencing and any drugs you may be taking.
* Blood (about 2 tablespoons) will be drawn for routine tests.

On Day 5 of Cycle 1 and Days 1 and 5 of Cycle 2, before you receive any of the study drugs, blood (about 2 teaspoons each time) will be drawn to test for CIMP, a chemical "marker" in the blood that may be related to how the drug may affect the cancer.

After every 3 cycles (Cycles 4, 7, 10 and so on), you will have a CT or MRI scan of the chest, abdomen, and/or pelvis to check the status of the disease.

Length of Study:

You may continue to take the study drugs for as long as you are benefitting. You will be taken off the study drugs if the disease gets worse, you experience any intolerable side effects, or if the study doctor thinks it is in your best interest to stop taking the study drugs.

If you chose to stop your participation in this study at any time, you should tell the study doctor or study staff right away. They will make sure that proper procedures are followed and a final visit is made for your safety.

End-of-Treatment Visit:

Within 10 days after your study treatment ends for any reason, you will return to the clinic and the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight and vital signs.
* You will have a neurosensory assessment.
* Your performance status will be recorded.
* You will have a CT scan or MRI scan of the chest, abdomen, and/or pelvis to check the status of the disease.
* You will be asked about any symptoms and/or side effects you may be experiencing and any drugs you may be taking.
* Blood (about 2 tablespoons) will be drawn for routine tests.

Follow-Up:

The study doctor and study staff will follow your health status for the first 30 days after you stop taking the study drugs to check if you are experiencing any treatment-related side effects. The follow-up will be done during your regularly scheduled routine clinic visits and/or by phone call, which should last about 5 minutes.

If you continue to experience any treatment-related side effects after the 30 days of follow-up, the study staff will continue to follow up with you during your regularly scheduled clinic visits until the side effects have gotten better or become stable.

Long-Term Follow-Up:

Every 3 months after the end-of-treatment visit, the study staff will contact you by phone or email to check on how you are doing. If you are contacted by phone, the call should last about 5 minutes. Your medical records may also be reviewed.

This is an investigational study. Azacitidine is FDA approved and commercially available for myelodysplastic syndrome (MDS - a blood disease that often leads to cancer). Its use in colorectal cancer is investigational.

Oxaliplatin and capecitabine are both FDA approved and commercially available as treatment for colorectal cancer.

The use of azacitidine, oxaliplatin, and capecitabine in combination is investigational.

Up to 54 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Phase I: Patient must have histologically or cytologically confirmed colorectal adenocarcinoma with metastatic disease documented on diagnostic imaging studies. Disease may be measurable or non-measurable as per RECIST version 1.1.
2. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
3. For patients on full-dose low-molecular weight anticoagulation, no active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or know varices) is allowed.
4. Serum bilirubin levels </= 1.5 times the upper limit of the normal range for the laboratory (ULN)
5. Serum aspartate aminotransferase (AST) or serum alanine aminotransferase (ALT) levels </= 2.5 x ULN and </= 5 x ULN in patients with liver metastases
6. Serum creatinine levels </= 1.5 x ULN
7. Absolute neutrophil count of >/=1,500/mm^3 (ie, >/=1.5 x 10^9/L by International Units [IU]).
8. Platelet count >/=100,000/mm^3 (IU: ≥100 x 10^9/L).
9. Hemoglobin value of >/=9.0 g/dL.
10. No limit to number of prior therapies.
11. Women of childbearing potential must have a negative serum pregnancy test and must be advised to avoid becoming pregnant. Men should be advised to not father a child while receiving treatment. Sexually active women of childbearing potential and men must use an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized.
12. Patient must be refractory to treatment with 5-FU (either intravenous 5-FU or as the oral prodrug, capecitabine) and oxaliplatin, defined as previous clinical or radiographic progression on or within 3 months of treatment with 5-FU and oxaliplatin. There is no limit to the number of prior lines of therapy.
13. Phase II: Patient must have histologically or cytologically confirmed colorectal adenocarcinoma with measurable metastatic disease documented on diagnostic imaging studies by RECIST version 1.1 criteria
14. Phase II: Patient must be known to have CpG island methylator phenotype.

Exclusion Criteria:

1. Patients with known brain metastases or carcinomatous meningitis
2. Patients unable to swallow oral medications or with gastrointestinal disorders that might interfere with proper absorption of oral drugs.
3. Known dihydropyrimidine (DPD) deficiency
4. Grade 3 or more peripheral neuropathy
5. Chemotherapy or any other investigational agents within 14 days of first receipt of study treatment, or major surgery within 28 days of first receipt of study treatment, or palliative radiation within 7 days of first receipt of study treatment.
6. Concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study such as unstable angina, myocardial infarction within 6 months, unstable symptomatic arrhythmia, uncontrolled diabetes, serious active or uncontrolled infection.
7. Known or suspected hypersensitivity to azacitidine or mannitol
8. Pregnant or breast feeding
9. Because of the interaction between coumadin and capecitabine patients taking therapeutic doses of coumarin-derivative anticoagulants, are not eligible. Low-dose Coumadin (e.g. 1 mg PO per day) in patients with in-dwelling venous access devices is allowed but increased frequency of international normalized ratio (INR) monitoring is recommended.
10. Interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Overman, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: August 2010 to August 2013. All recruitment done at The University of Texas MD Anderson Cancer Center.
Groups:
- Phase I: Starting Dose: Dose Escalation of Azacitidine + CAPOX (Capecitabine, Oxaliplatin)
  Of 21 day cycle, starting dose Azacitidine 75 mg/m2/day subcutaneously on Days 1-5; Capecitabine 1500 mg/m2/day by mouth twice daily in divided doses on Days 1-14; and Oxaliplatin starting dose 90 mg/m2 by vein on Day 2.
- Phase I: Highest Dose Level: Subcutaneous Azacitidine 75 mg/m2/day days 1 to 5, intravenous Oxaliplatin 110 mg/m2 day 2, and oral capecitabine 1500 mg/m2 divided twice daily for 2 weeks every three weeks
- Phase II: MTD of Azacitidine + CAPOX
  Of a 21 day cycle, Azacitidine MTD (Highest tolerable dose of combination azacitidine with CAPOX found in Phase I); Capecitabine 1500 mg/m2/day by mouth twice daily in divided doses on Days 1-14; and Oxaliplatin starting dose 90 mg/m2 by vein on Day 2.
Period: Overall Study
Arm/Group | Phase I: Starting Dose | Phase I: Highest Dose Level | Phase II
Started | 3 | 12 | 11
Completed | 2 | 12 | 11
Not Completed | 1 | 0 | 0
Not completed — Early Progression | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: Starting Dose | Phase I: Highest Dose Level | Phase II | Total
Number analyzed (Participants) | 3 | 12 | 11 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 9 | 7 | 18
  >=65 years | 1 | 3 | 4 | 8
Age, Continuous [Mean (Full Range); unit: years] | 59 [51 to 68] | 56 [33 to 73] | 61 [48 to 75] | 59 [33 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 4 | 11
  Male | 2 | 6 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 3 | 10 | 11 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 3
  White | 2 | 8 | 9 | 19
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 12 | 11 | 26

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Azacitidine, and Capecitabine and Oxaliplatin (CAPOX)
Description: Dose just below the one at which ≥ 1/3 of subjects experience a dose limiting toxicity (DLT) considered the MTD.
Time Frame: Up to 3 weeks from the first dose
Measure: Number; unit: mg/m^2
Groups:
- Azacitidine+CAPOX (Capecitabine, Oxaliplatin): Subcutaneous Azacitidine 75 mg/m2/day days 1 to 5, intravenous Oxaliplatin 110 mg/m2 day 2, and oral capecitabine 1500 mg/m2 divided twice daily for 2 weeks every three weeks
Arm/Group | Azacitidine+CAPOX (Capecitabine, Oxaliplatin)
Number analyzed (Participants) | 26
mg/m^2
  Azacitidine | 75
  Oxaliplatin | 110
  Capecitabine | 1500

2. Secondary Outcome: Response Rate of Azacitidine, and Capecitabine and Oxaliplatin (CAPOX)
Description: Per Response Evaluation Criteria in solid Tumors Criteria (RECISTv1.0) for target lesions and assessed by CT or MRI: Partial Response (PR), >= 30%decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither PD nor PR, the sum of the longest diameters no change or increase by <20% from baseline or from nadir (smallest sum on treatment); Progressive Disease (PD), the sum of the longest diameters increases by>= 20% from nadir (smallest sum on treatment). For non-target lesions assessed by CT or MRI: Stable Disease (SD), Persistence of >=1 non-target lesion; Progressive Disease (PD), Enlargement of non-target lesions and/or appearance of new lesions.
Time Frame: After 9 weeks (three, 21 day cycles)
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Starting Dose | Phase I: Highest Dose Level | Phase II
Number analyzed (Participants) | 3 | 12 | 11
Participants
  NA (Early Progression) | 1 | 0 | 0
  PD (Progression Disease) | 1 | 6 | 1
  SD (Stable Disease) | 1 | 6 | 10

ADVERSE EVENTS:
Time Frame: Adverse event data collected from baseline, during active 21 day cycle treatment and for 30 days after the last dose of study drug
Arm/Group | Phase I: Starting Dose | Phase I: Highest Dose Level | Phase II
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/12 | 1/11
Other Adverse Events (participants affected / at risk) | 2/3 | 12/12 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Starting Dose (N=3) | Phase I: Highest Dose Level (N=12) | Phase II (N=11)
Nausea (Gastrointestinal disorders) | 0 | 2 | 1
Vomitting (Gastrointestinal disorders) | 0 | 1 | 1
Pain-pelvis (General disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Starting Dose (N=3) | Phase I: Highest Dose Level (N=12) | Phase II (N=11)
Nausea (Gastrointestinal disorders) | 1 | 9 | 8
Vomiting (Gastrointestinal disorders) | 1 | 5 | 6
Neuropathy Sensory (Nervous system disorders) | 1 | 1 | 6
Neutrophils (Blood and lymphatic system disorders) | 2 | 7 | 7
Anorexia (Gastrointestinal disorders) | 1 | 6 | 6
Diarrhea (Gastrointestinal disorders) | 1 | 6 | 5
Flatulence (Gastrointestinal disorders) | 1 | 1 | 0
Fatigue (General disorders) | 1 | 9 | 9
Platelet (Blood and lymphatic system disorders) | 0 | 5 | 8
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Sodium, Serum-low (Metabolism and nutrition disorders) | 0 | 0 | 1
Phosphase, Serum-low (Metabolism and nutrition disorders) | 0 | 1 | 0
Potassium, Serum-low (Metabolism and nutrition disorders) | 0 | 2 | 3
Magnesium, Serum-low (Metabolism and nutrition disorders) | 0 | 2 | 3
Potassium, Serum-High (Metabolism and nutrition disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 2
Leukocytes (Blood and lymphatic system disorders) | 0 | 2 | 1
Fever (General disorders) | 0 | 3 | 1
Alkaline Phasphatase (Metabolism and nutrition disorders) | 0 | 0 | 3
ALT (Metabolism and nutrition disorders) | 0 | 2 | 4
AST (Metabolism and nutrition disorders) | 0 | 7 | 4
Hemoglobin (Blood and lymphatic system disorders) | 0 | 7 | 7
Neurology Other (Nervous system disorders) | 0 | 1 | 1
Pain Other-injection site (General disorders) | 0 | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Glucose, Serum-high (Metabolism and nutrition disorders) | 0 | 1 | 0
Taste Alteration (Gastrointestinal disorders) | 0 | 1 | 4
Hypersensitivity (Immune system disorders) | 0 | 2 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 0 | 3 | 10
Flu-like Syndrome (Immune system disorders) | 0 | 3 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
UTI (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 1 | 0
hemorrhage, pulmonary-hemoptysis (Blood and lymphatic system disorders) | 0 | 1 | 0
Sweating (General disorders) | 0 | 1 | 0
Pain-Muscle (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain - Joint (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Edema-Limbs (Blood and lymphatic system disorders) | 0 | 1 | 0
Rash; Hand-Foot Skin Reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Weight Loss (General disorders) | 0 | 1 | 2
Dizziness (Nervous system disorders) | 0 | 2 | 0
Dehydration (Gastrointestinal disorders) | 0 | 2 | 3
Pulmonary-Other Throat Tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bilirubin (Blood and lymphatic system disorders) | 0 | 2 | 5
Rash Desquamation (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Vision-Blurred (Eye disorders) | 0 | 1 | 1
Hemorrhage-Other (Blood and lymphatic system disorders) | 0 | 0 | 1
Pain-Abdomen NOS (Gastrointestinal disorders) | 0 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Hypertension (Cardiac disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Ileus, GI-small Intestine (Gastrointestinal disorders) | 0 | 0 | 1
Wartering Eye (Eye disorders) | 0 | 0 | 1
Ocular/Visual-other (Eye disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes